CLINICAL TRIAL: NCT03276793
Title: Using Human Brain Connectivity to Identify the Causal Neuroanatomical Substrate of Depression Symptoms
Brief Title: Brain Connectivity in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Butler Hospital (Other); Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael D. Fox, M.D.,Ph.D., Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021P000335; R01MH113929 (NIH)
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2025-04-21 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI and behavioral assessment for patients receiving TMS (Experimental): Subjects will undergo an hour-long MRI scanning session, a marking for the site of planned clinical TMS stimulation and a behavioral testing battery before and after their TMS treatment course.
  Interventions: Other: MRI scan; Behavioral: Behavioral testing

INTERVENTIONS:
Other: MRI scan — Patients will undergo an MRI scan
Behavioral: Behavioral testing — Patients will complete a series of cognitive tasks

SUMMARY:
This study originally included 140 subjects with medication-refractory depression undergoing 10 Hz transcranial magnetic stimulation (10Hz-TMS) to the left dorsal lateral prefrontal cortex (DLPFC), with the goal of having 60 completers with good quality data. Subjects were recruited from the TMS clinics at Beth Israel Deaconess Medical Center, Brigham & Women's Hospital, and Butler Hospital. Subjects underwent an hour-long MRI scanning session, an optional DNA-sample collection, up to three 20 minute neuronavigation sessions for marking the site of TMS stimulation, questionnaires, and a behavioral testing battery before and after their TMS treatment course. The task battery included the Emotion Conflict Resolution (ECR) task, Multi-Source Interference Task (MSIT), War Game (Gambling) task, and Associative Learning with Reversal task. Subjects' scores on the Quick Inventory of Depressive Symptomatology (QIDS) and Beck Depression Inventory (BDI) were assessed before and after the TMS course. MRI data was utilized to identify brain regions whose connectivity to the stimulation site co-varies with the aforementioned measures of symptom improvement. This was the only study group until August 30, 2022, and the primary outcome was analyzed for the 10Hz-TMS group.

Due to changes in clinical standard of care from 10Hz-TMS to a newer version of TMS termed intermittent theta burst (iTBS), in September 2022 a second group was added to include patients receiving this new form of TMS. This second group included another 100 patients with medication-refractory depression undergoing iTBS to the left dorsal lateral prefrontal cortex (DLPFC), with the intent to have 80 completers. Massachusetts General Hospital was added as a data collection site in lieu of Butler Hospital. Subjects will undergo an hour-long MRI scanning session, up to three 20 minute neuronavigation sessions for marking the site of TMS stimulation, questionnaires, and a behavioral testing battery before and after their TMS treatment course. The task battery will included the Emotion Conflict Resolution (ECR) task, Multi-Source Interference Task (MSIT), Penn Emotion Recognition Test, the Suicide/Death Implicit Association Test, and Associative Learning with Reversal task. Subjects' scores on the Beck Depression Inventory (BDI) were assessed before and after the TMS course. MRI data will be utilized to identify brain regions whose connectivity to the stimulation site co-varies with the aforementioned measures of symptom improvement.

Due to a higher dropout rate than anticipated, in March of 2025 an amendment was added to include an additional 20 subjects in the second group's enrollment goal to increase the likelihood of achieving 80 completers.

DETAILED DESCRIPTION:
This study was originally approved by the Beth Israel Deaconess Medical Center (BIDMC) Institutional Review Board (IRB) with Butler Hospital as a relying site. The study was transferred to the Mass General Brigham (MGB) IRB in 2020 when Dr. Fox (lead PI) moved to Brigham and Women's Hospital (BWH). Butler Hospital continued to enroll subjects, relying on the MGB IRB for regulatory oversight, while BIDMC stopped enrolling subjects. A Data Usage Agreement was established between BIDMC and BWH, and all previously collected Data was de-identified and sent to BWH. The protocol at BIDMC will remain active but not enrolling until all the de-identified data has been sent to BWH.

In Sept 2022, with the launch of the second iTBS group, Massachusetts General Hospital replaced Butler Hospital as the secondary enrollment site, while enrollment continued at Brigham and Women's Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged 18 or older
3. Have previously received or will once daily TMS treatment to the left dorsolateral prefrontal cortex at the Center for Brain Circuit Therapeutics at Brigham and Women's Hospital, or at Massachusetts General Hospital for treatment of medication resistant depression

Exclusion Criteria:

1. Presence of a significant neurologic disorder (i.e. Parkinson's Disease, stroke, Alzheimer's Disease, tumor, multiple sclerosis, epilepsy) or other significant active medical problems which may impact treatment or safety. Of note, many of these are also contraindications to receiving TMS and these patients would not be enrolled in the clinical treatment program. Because these diagnoses, their significance, and the extent to which they are an active issue can be subjective, each of these exclusions (1-3) will be reviewed by the PI or study physician
2. Lack of response to an adequate trial of electroconvulsive therapy (ECT) or any ECT in the preceding 3 months
3. Prior adequate trial of TMS treatment in the last 12 months
4. Positive MRI screen that would preclude the subject from undergoing magnetic resonance imaging. These include, but are not limited to any of the following:

   1. Known metal in the head (such as a surgical aneurysm clip), or a history of prior neurosurgical procedures
   2. Ferromagnetic bioimplants activated by any electronic, mechanical or magnetic means such as: cochlear implants, pacemakers, medication pumps, vagal stimulators, deep brain stimulators, neurostimulators, biostimulators, or ventriculo-peritoneal shunts
   3. Subjects who have or might have bullet fragments or other metal fragments (veterans or workers exposed to metal in their work environment)
   4. Subjects with metallic paint (e.g. color contact lenses, tattoos, metallic eyeliner)
   5. Subjects expressing significant anxiety or claustrophobia about being in the magnet.
5. Subjects that cannot adhere to the experimental protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of repetitive Transcranial Magnetic Stimulation (rTMS) clinical response | 1 year after study completion
  Connectivity between each patient's stimulation site and the subgenual cingulate will be used to predict clinical response to rTMS in the first group (data collected starting in 2017).
Prediction of intermittent theta burst stimulation (iTBS) clinical response | 1 year after study completion
  Normative connectivity of each patient's stimulation site to a previously-published "depression network" (Siddiqi et al., Nat Hum Behav 2021) will be used to predict clinical response to iTBS in the second group added in September 2022.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Butler Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khosravani S, Palm ST, Drew W, Frandsen SB, Lin C, Tirrell E, Hindley L, Schineller M, Garimella A, Chiulli N, Lawson D, Jones E, Press DZ, Stern AP, Brown JC, Barbour TA, Taylor JJ, Carpenter LL, Siddiqi SH, Fox MD. Predictive value of subgenual cingulate normative connectivity to TMS treatment site for antidepressant response in routine clinical practice: a prospective, multisite cohort study. Mol Psychiatry. 2026 Feb;31(2):689-700. doi: 10.1038/s41380-025-03153-3. Epub 2025 Aug 22. PMID 40847007